CLINICAL TRIAL: NCT03525548
Title: A Phase 3, Randomized, Double-blind, Controlled Study Evaluating the Efficacy and Safety of VX-445 Combination Therapy in Subjects With Cystic Fibrosis Who Are Homozygous for the F508del Mutation (F/F)
Brief Title: A Study of VX-445 Combination Therapy in CF Subjects Homozygous for F508del (F/F)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX17-445-103; 2018-000184-89 (EudraCT Number)
Expanded Access: NCT04058210 (Approved for marketing)
Record Dates: First submitted 2018-05-02; First posted 2018-05-15 (Actual); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor; tezacaftor, ivacaftor drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TEZ/IVA (Active Comparator): Following a run-in period of 4 weeks with Tezacaftor (TEZ)/Ivacaftor (IVA), participants received TEZ 100 milligram (mg)/IVA 150 mg as fixed-dose combination (FDC) tablet in the morning and IVA 150 mg as mono tablet in the evening for 4 weeks in the triple combination (TC) treatment period.
  Interventions: Drug: TEZ/IVA; Drug: IVA; Drug: Placebo
- VX-445/TEZ/IVA TC (Experimental): Following a run-in period of 4 weeks with TEZ/IVA, participants received VX-445 200 mg/TEZ 100 mg/IVA 150 mg as FDC tablets in the morning and IVA 150 mg as mono tablet in the evening for 4 weeks in the TC treatment period.
  Interventions: Drug: VX-445/TEZ/IVA; Drug: IVA; Drug: Placebo

INTERVENTIONS:
Drug: VX-445/TEZ/IVA — Participants received VX-445/TEZ/IVA orally once daily in the morning.
  Other Names: VX-445/VX-661/VX-770; VX-445/tezacaftor/ivacaftor
  Arms: VX-445/TEZ/IVA TC
Drug: TEZ/IVA — Participants received TEZ/IVA orally once daily in the morning.
  Other Names: VX-661/VX-770; tezacaftor/ivacaftor
  Arms: TEZ/IVA
Drug: IVA — Participants received IVA orally once daily in the evening.
  Other Names: VX-770; ivacaftor
Drug: Placebo — Participants received placebo matched to VX-445/TEZ/IVA orally once daily in the morning.
  Arms: TEZ/IVA
Drug: Placebo — Participants received placebo matched TEZ/IVA orally once daily in the morning.
  Arms: VX-445/TEZ/IVA TC

SUMMARY:
This study will evaluate the efficacy of VX-445 in triple combination (TC) with tezacaftor (TEZ) and ivacaftor (IVA) in subjects with cystic fibrosis (CF) who are homozygous for the F508del mutation (F/F)

ELIGIBILITY:
Key Inclusion Criteria:

* Homozygous for the F508del mutation (F/F)
* Forced expiratory volume in 1 second (FEV1) value ≥40% and ≤90% of predicted mean for age, sex, and height

Key Exclusion Criteria:

* Clinically significant cirrhosis with or without portal hypertension
* Lung infection with organisms associated with a more rapid decline in pulmonary status
* Solid organ or hematological transplantation

Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (44):
- United States (28):
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Miller Children's Hospital/ Long Beach Memorial, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - National Jewish Health, Denver, Colorado
  - Joe DiMaggio Cystic Fibrosis & Pulmonary Center/ Joe DiMaggio Children's Hospital/ Memorial Regional Hospital, Hollywood, Florida
  - Central Florida Pulmonary Group, PA, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Tampa General Hospital Cardiac and Lung Transplant Clinic, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Saint Francis Medical Center/ Children's Hospital of Illinoise/OSF, Peoria, Illinois
  - Tulane Medical Center, New Orleans, Louisiana
  - Massachusetts General Hospital Cystic Fibrosis Center Clinical Research Center, Boston, Massachusetts
  - Harper University Hospital, Detroit, Michigan
  - New York Medical College, Valhalla, New York
  - UNC Marisco Clinical Research Center, Chapel Hill, North Carolina
  - Rainbow Babies and Children's Hospital/University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/ Toledo Children's Hospital/ Pediatric Pulmonary & Cystic Fibrosis Center, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Vermont Lung Center, Colchester, Vermont
  - University of Virginia Primary Care Center, Charlottesville, Virginia
  - West Virginia University, Morgantown, West Virginia
- Belgium (5):
  - Cliniques Universitaires de Bruxelles Hopital Erasme, Brussels
  - Universitair Ziekenhuis Brussel - Campus Jette, Brussels
  - UZ Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- Netherlands (5):
  - Academic Medical Center, Amsterdam
  - University Medical Center, Utrecht, Department of Pulmonology and Tuberculosis, Heidelberglaan
  - UMC St. Radboud, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - HagaZiekenhuis van den Haag, The Hague
- United Kingdom (6):
  - The Royal Belfast Hospital for Sick Children, Belfast
  - Heart of England NHS Foundation Trust, Birmingham Heartlands Hospital, Birmingham
  - Royal Devon and Exeter NHS Foundation Trust, Royal Devon and Exeter Hospital, Exeter
  - Leeds General Infirmary, Leeds
  - King's College Hospital, London
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Heijerman HGM, McKone EF, Downey DG, Van Braeckel E, Rowe SM, Tullis E, Mall MA, Welter JJ, Ramsey BW, McKee CM, Marigowda G, Moskowitz SM, Waltz D, Sosnay PR, Simard C, Ahluwalia N, Xuan F, Zhang Y, Taylor-Cousar JL, McCoy KS; VX17-445-103 Trial Group. Efficacy and safety of the elexacaftor plus tezacaftor plus ivacaftor combination regimen in people with cystic fibrosis homozygous for the F508del mutation: a double-blind, randomised, phase 3 trial. Lancet. 2019 Nov 23;394(10212):1940-1948. doi: 10.1016/S0140-6736(19)32597-8. Epub 2019 Oct 31. PMID 31679946

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 113 participants were enrolled in the study, of which 6 participants were included in the run-in period but were not dosed in TC treatment period. Results are presented for 107 participants dosed in the TC treatment period.
Pre-assignment Details: This study was conducted in participants with cystic fibrosis (CF) aged 12 years or older.
Groups:
- TEZ/IVA: Following a run-in period of 4 weeks with TEZ/IVA, participants received TEZ 100 mg/IVA 150 mg as FDC tablet in the morning and IVA 150 mg as mono tablet in the evening for 4 weeks in the TC treatment period.
Period: Overall Study
Arm/Group | TEZ/IVA | VX-445/TEZ/IVA TC
Started | 52 | 55
Completed | 52 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TEZ/IVA | VX-445/TEZ/IVA TC | Total
Number analyzed (Participants) | 52 | 55 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.9 (10.8) | 28.8 (11.5) | 28.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 31 | 59
  Male | 24 | 24 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 49 | 52 | 101
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 52 | 54 | 106
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) [Mean (Standard Deviation); unit: percentage points] — FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
  percentage points | 60.2 (14.4) | 61.6 (15.4) | 60.9 (14.9)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline at Week 4
Population: Full analysis set (FAS) included all randomized participants who carried the intended CF transmembrane conductance regulator gene (CFTR) allele mutation and received at least 1 dose of study drug in the TC Treatment Period.
Measure: Least Squares Mean (Standard Error); unit: percentage points
Arm/Group | TEZ/IVA | VX-445/TEZ/IVA TC
Number analyzed (Participants) | 52 | 55
percentage points | 0.4 (0.9) | 10.4 (0.9)
Statistical Analysis 1: Comparison: TEZ/IVA vs VX-445/TEZ/IVA TC; Test type: Superiority; p < 0.0001, Mixed-effects model for repeated measure; Least squares (LS) mean difference = 10, 95% CI 2-sided [7.4 to 12.6]

2. Secondary Outcome: Absolute Change in Sweat Chloride (SwCl)
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline at Week 4
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | TEZ/IVA | VX-445/TEZ/IVA TC
Number analyzed (Participants) | 52 | 55
millimole per liter (mmol/L) | 1.7 (1.8) | -43.4 (1.7)
Statistical Analysis 1: Comparison: TEZ/IVA vs VX-445/TEZ/IVA TC; Test type: Superiority; p < 0.0001, Mixed-effects model for repeated measure; LS mean difference = -45.1, 95% CI 2-sided [-50.1 to -40.1]

3. Secondary Outcome: Absolute Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicate fewer symptoms and better health-related quality of life.
Time Frame: From Baseline at Week 4
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TEZ/IVA | VX-445/TEZ/IVA TC
Number analyzed (Participants) | 52 | 55
units on a scale | -1.4 (2.0) | 16.0 (2.0)
Statistical Analysis 1: Comparison: TEZ/IVA vs VX-445/TEZ/IVA TC; Test type: Superiority; p < 0.0001, Mixed-effects model for repeated measure; LS mean difference = 17.4, 95% CI 2-sided [11.8 to 23.0]

4. Secondary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: From first dose of study drug in TC treatment period up to 28 days after last dose of study drug or to the completion of study participation date, whichever occurs first (up to Week 8)
Population: Safety set included all participants who received at least 1 dose of study drug in the TC treatment period.
Measure: Number; unit: participants
Arm/Group | TEZ/IVA | VX-445/TEZ/IVA TC
Number analyzed (Participants) | 52 | 55
participants
  Participants with AEs | 33 | 32
  Participants with SAEs | 1 | 2

5. Secondary Outcome: Observed Pre-Dose Concentration (Ctrough) of VX-445, TEZ, TEZ Metabolite (M1-TEZ), and IVA
Time Frame: Day 1 and Week 4
Population: Pharmacokinetic analysis set included all participants who received at least 1 dose of study drug in the TC treatment period. Here "Number analyzed" signifies those participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | TEZ/IVA | VX-445/TEZ/IVA TC
Number analyzed (Participants) | 52 | 55
microgram per milliliter (mcg/mL)
  VX-445: Day 1: number analyzed (Participants) | 0 | 55
  VX-445: Day 1 |  | NA (NA) — Data was not reported at the specified time point as all the observations were below the limit of quantitation.
  VX-445: Week 4: number analyzed (Participants) | 0 | 54
  VX-445: Week 4 |  | 4.84 (2.59)
  TEZ: Day 1: number analyzed (Participants) | 50 | 55
  TEZ: Day 1 | 1.71 (0.942) | 1.60 (1.03)
  TEZ: Week 4 | 1.48 (0.829) | 1.89 (0.974)
  M1-TEZ: Day 1: number analyzed (Participants) | 50 | 55
  M1-TEZ: Day 1 | 4.84 (1.71) | 4.76 (1.78)
  M1-TEZ: Week 4 | 4.86 (1.74) | 5.28 (2.04)
  IVA: Day 1: number analyzed (Participants) | 50 | 55
  IVA: Day 1 | 0.652 (0.399) | 0.598 (0.428)
  IVA: Week 4 | 0.530 (0.297) | 0.652 (0.542)

ADVERSE EVENTS:
Time Frame: From first dose of study drug in TC treatment period up to 28 days after last dose of study drug or to the completion of study participation date, whichever occurs first (up to Week 8)
Arm/Group | TEZ/IVA | VX-445/TEZ/IVA TC
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/55
Serious Adverse Events (participants affected / at risk) | 1/52 | 2/55
Other Adverse Events (participants affected / at risk) | 25/52 | 24/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TEZ/IVA (N=52) | VX-445/TEZ/IVA TC (N=55)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TEZ/IVA (N=52) | VX-445/TEZ/IVA TC (N=55)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Nasopharyngitis (Infections and infestations) | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 2 | 4
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 3 | 1
Headache (Nervous system disorders) | 4 | 3
Fatigue (General disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/48/NCT03525548/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/48/NCT03525548/SAP_001.pdf